CLINICAL TRIAL: NCT01332643
Title: Comparison of Single Embryo Transfer With and Without Previous Analysis of All Chromosome Abnormalities Using Microarrays
Brief Title: Preimplantation Genetic Diagnosis (PGD) by Array Comparative Genome Hybridization (CGH) and Blastocyst Biopsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough patients enrolling
Sponsor: Reprogenetics (Industry)
Collaborators: Reprogenetics Lationoamerica S.A.C, Lima, Peru (Unknown); Pranor S.R.L., Lima, Peru (Unknown); Yale University (Other); McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reprogenetics-02
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Infertility; Miscarriage
Keywords: Preimplantation Genetic Diagnosis; recurrent pregnancy loss; infertility; genetic screening; trisomy 21; Down syndrome
MeSH Terms: conditions — Infertility; Abortion, Spontaneous; Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test (Active Comparator): The test group will consist of patients undergoing blastocyst biopsy followed by vitrification (embryo freezing), and in which the biopsied cells will be analyzed with a comprehensive chromosome analysis technique (array Comparative Genome hybridization or aCGH) and only one chromosomally normal embryo will be replaced in a thawed cycle.
  Interventions: Genetic: Preimplantation Genetic Diagnosis
- control (No Intervention): The control group will consist of patients in which one embryo will be replaced on day 5 based on morphological and developmental characteristics, and the other embryos reaching blastocyst stage will be vitrified. If patient does not become pregnant, successive embryo transfers of frozen embryos will be performed, but not as part of the study.

INTERVENTIONS:
Genetic: Preimplantation Genetic Diagnosis — All embryos in the test group reaching blastocyst stage will undergo embryo biopsy of 3-10 trophectoderm cells. The cells will be analyzed by array CGH to detect the presence or not of chromosome abnormalities. The embryos will be vitrified and those classified by array CGH as normal, thawed for replacement.
  Other Names: array CGH from Bluegnome, UK
  Arms: Test

SUMMARY:
This study evaluates the effect of single embryo transfer (SET) with and without array CGH for the evaluation of the complete chromosome complement of the blastocyst. Patients will be allocated at random into two groups. The control group will consist of patients in which one embryo will be replaced on day 5 based on morphological and developmental characteristics, and the other embryos reaching blastocyst stage will be vitrified. The test group will consist of patients undergoing embryo biopsy at the blastocyst stage (day 5 of development, embryo freezing, and analysis of the biopsied cells with a comprehensive chromosome analysis technique (array Comparative Genome hybridization or aCGH). Only a chromosomally normal blastocyst will be replaced in a thawed cycle. Inclusion and exclusion criteria are described in the study population section.

DETAILED DESCRIPTION:
Rational for the study:

The goal of this study is to determine if the strategy employed for the Test group can solve two major problems in ART, one the still low implantation rate in women of advanced maternal age, and two the frequent occurrence of multiple pregnancies resulting from solving the first problem by replacing too many embryos.

Preimplantation Genetic Diagnosis (PGD) has been proposed as a potential means to achieve these goals, but so far, the results with day 3 biopsy and FISH analysis of 5-12 chromosomes has produced contradictory results, the difference between studies being explained by technical differences (Munne et al. 2010). Three technical developments have recently occurred that can change dramatically the efficacy of PGD. One, blastocyst laser assisted biopsy, which seems less detrimental than cleavage stage biopsy; Two, vitrification of embryos which allows those blastocysts to be frozen with little or no loss of viability, and three, chromosome comprehensive screening techniques, such as array CGH (Gutierrez-Mateo et al. 2011) which allow for the detection of all chromosome abnormalities.

Preliminary data from our center indicates that the technique to be used, an improvement on our prior technique CGH, will result in a very significant improvement in implantation rates and a reduction in miscarriage rates, thus justifying the use of single embryo transfer in this set up.

Supportive Preliminary Research:

In a recent study, the investigators observed a 1.6 fold increase (p < 0.001) in implantation rate when aCGH was applied to blastocyst embryos (Schoolcraft et al. 2010). The test group used CGH, an older and less sensitive iteration of the technique to be used in the proposed study - array CGH. Array CGH has a 6 megabase resolution and screens for 30% of all DNA bases (compared to 0.1% of SNP arrays). With array CGH the false positive and false negative rate is 0% when biopsying blastocysts, and 3% when biopsying day 3 embryos (Gutierrez Mateo et al, 2011). Based on our preliminary data, patients with 5 or more day 3 embryos and less than 43 years of age are the most likely to benefit from PGD, since they produce enough embryos and enough normal embryos so a selection technique, like PGD could chose them and improve their reproductive odds.

Also our PGD preliminary data shows a < 10% of embryo demise after implantation for a population 38 of age (expected would be about 28%).

Study Hypothesis The investigators foresee a significant increase in implantation rates in the Test group compared to the Control group. The investigators calculated that 60 patients in each arm would be needed to achieve a significant increase in implantation rates (p < 0.05) with a power of 80%, based on a comparative study in which the investigators observed a 1.6 fold increase in implantation rate (Schoolcraft et al. 2010).

Study population, interventions:

see below.

ELIGIBILITY:
Inclusion Criteria:

* Couples with women 30-42 years of age
* Follicle Stimulating Hormone (FSH) level <11IU/L on day 3 of cycle.

Exclusion Criteria:

* TESA and TESE patients
* Couples' carriers of chromosomal or genetic diseases
* Couples that produce less than eight antral follicles on day 2-4 of cycle
* Patients will be excluded if they produce no blastocysts by day 5

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | three weeks after embryo replacement
  number of embryos implanted divided by number of embryos replaced. An embryo implanted is measured as a fetal sac by ultrasound observation.

SECONDARY OUTCOMES:
miscarriage rate | up to the end of second trimester
  lost pregnancies, defined as pregnancies with an observed fetal sac that did not progressed to third trimester.
Pregnancy rate per transfer | three weeks after implantation
  pregnancy defined as the presence of a fetal sac. Pregancy rate per transfer defined as pregnancies divided by patients with a replacement of embryos.
Pregnancy rate per retrieval | three weeks after transfer
  pregnancy defined as the presence of a fetal sac. Pregancy rate per retrieval defined as pregnancies divided by patients with an egg retrieval.
live birth rate | 1 year after embryo transfer
  pregnancies that arrive to term divided by procedures with an egg retreival.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Munne, PhD, Principal Investigator — Reprogenetics
Locations (1):
- Pranor, Lima, Lima Province, Peru

REFERENCES:
- [Background] Gutierrez-Mateo C, Colls P, Sanchez-Garcia J, Escudero T, Prates R, Ketterson K, Wells D, Munne S. Validation of microarray comparative genomic hybridization for comprehensive chromosome analysis of embryos. Fertil Steril. 2011 Mar 1;95(3):953-8. doi: 10.1016/j.fertnstert.2010.09.010. Epub 2010 Oct 25. PMID 20971462
- [Background] Schoolcraft WB, Fragouli E, Stevens J, Munne S, Katz-Jaffe MG, Wells D. Clinical application of comprehensive chromosomal screening at the blastocyst stage. Fertil Steril. 2010 Oct;94(5):1700-6. doi: 10.1016/j.fertnstert.2009.10.015. Epub 2009 Nov 25. PMID 19939370
- [Background] Munne S, Wells D, Cohen J. Technology requirements for preimplantation genetic diagnosis to improve assisted reproduction outcomes. Fertil Steril. 2010 Jul;94(2):408-30. doi: 10.1016/j.fertnstert.2009.02.091. Epub 2009 May 5. PMID 19409550